CLINICAL TRIAL: NCT06920641
Title: Effects of Tagatose on Glycemic Response and Gastrointestinal Microbiota: A Randomized, Placebo-Controlled, Double-Blind, Crossover Trial in Healthy Adults
Brief Title: Effects of Tagatose on Glycemic Response and Gastrointestinal Microbiota in Healthy Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-2413
Record Dates: First submitted 2025-03-25; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Glucose Intolerance; Microbial Colonization
Keywords: tagatose; prebiotic; fecal microbiota; glucose; insulin; gut health; glycemic control
MeSH Terms: conditions — Glucose Intolerance; Communicable Diseases; Insulin Resistance | interventions — tagatose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tagatose (Experimental): 10 grams tagatose
  Interventions: Other: Tagatose
- Placebo (Placebo Comparator): 10 grams sucrose
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Tagatose — Sachet containing 10g tagatose to be dissolved in 250ml water and taken once daily on Days 1-28 of a 4-week dosing period.
  (1 of 2 dosing periods separated by a 4-week washout)
  Arms: Tagatose
Other: Placebo — Sachet containing 10g sucrose to be dissolved in 250ml water and taken once daily on Days 1-28 of a 4-week dosing period.
  (1 of 2 dosing periods separated by a 4-week washout)
  Arms: Placebo

SUMMARY:
The primary objective of this clinical-trial is to determine, in subjects with impaired fasting glucose (IFG) and/or insulin resistance (IR), if tagatose meets the definition of a prebiotic, namely that consuming tagatose for 4 weeks selectively stimulates the selective growth of bacteria in the colon and is associated with a health benefit (oral glucose tolerance) when compared to consuming the control treatment (10g sucrose) for 4 weeks.

DETAILED DESCRIPTION:
Available evidence suggests that tagatose may act as a prebiotic compound. It has been hypothesized that undigested tagatose reaches the colon and is fermented by colonic bacteria, resulting in the production of short-chain fatty acids (SCFA) which stimulate GLP-1 secretion from colonic L-cells, which, in turn, improves glycemic control by increasing insulin sensitivity and insulin secretion. However, the fermentation of tagatose and subsequent effects have only been demonstrated in preclinical models, with limited clinical trials examining the effect of tagatose on glycemic control. Given the dearth of clinical evidence in humans supporting the ability of tagatose to be fermented in the colon and to improve glycemic control, the present study aims to explore if tagatose is selectively utilized by human gut microorganisms conferring a beneficial effect on glycemic control.

Thus, the investigators aim to recruit 55 healthy adults with impaired fasting glucose and/or hyperinsulinemia into a double-blind, randomized, controlled, clinical trial with a cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 18-50 years, inclusive
* BMI 20.0 to 34.9 kg/m², inclusive
* Fasting serum glucose <7.0 mmol/L
* Fasting serum glucose between 6.1 and 6.9 mmol/L (110 to 124 mg/dL), inclusive and/or fasting insulin >50th percentile (>43 pmol/L = >7.2 μU/mL)
* No history of diabetes mellitus
* Systolic blood pressure <160 mmHg and diastolic blood pressure <100 mmHg
* Agree not to change current dietary habits with the exception of the following: agreement to avoid foods/drinks with added probiotics, prebiotics, and/or postbiotics, fermented foods (e.g., yogurt, sauerkraut, kombucha), and dietary supplements containing fiber, probiotics, prebiotics, synbiotics, and/or postbiotics for at least 2 weeks before Week 0 (Day 1) and throughout the duration of their participation in the study
* Modified TAPS (tobacco, alcohol, prescription medications and other substances) tool responses are within allowable usage limits
* Ability to understand the study procedures and willing to provide informed consent to participate in the study
* Subjects must be eligible to receive income in Canada and be covered by a health insurance plan such as OHIP
* Subjects are willing to sign the informed consent prior to any procedures conducted

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Reported history of metabolic (including type 1 and type 2 diabetes mellitus), hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological, psychiatric disorders, or any other medical conditions that, in the judgment of the Principal Investigator, increase the risk to the subject or others or may affect results.
* Antibiotic use within 60 days before randomization
* Hospital admission for major trauma, or major medical or surgical event, as judged by the Principal Investigator, within 6 months of screening.
* Use of medications such as, but not limited to, hypoglycemic agents, GLP-I agonists, systemic steroids, antipsychotics, or any others that increase the risk to the subject or others or may affect results, as judged by the Principal Investigator.
* Current diagnosis or history of irritable bowel syndrome (IBS), inflammatory bowel disease (IBD, including ulcerative colitis and Crohn's disease), functional constipation (defined by the Rome IV diagnostic criteria 1-8, diarrhea (loose or watery stools for the last 3 months without abdominal pain or bothersome bloating in more than 25% of stools), celiac disease, lactose intolerance and/or malabsorption, gastroparesis, gastroenteritis, endometriosis, diverticulosis, gastric or duodenal ulcers, pancreatitis, or eating disorder; history of intestinal surgery (excluding appendectomy or herniorrhaphy), or history of bariatric surgery.
* Extreme dietary habits, including but not limited to intentional consumption of an extremely high fiber diet (e.g., >50g per day), gluten-free, low-carb, vegan, ketogenic, low FODMAP.
* Consumption of >2 sugar sweetened or artificially sweetened beverages (soda and juice) on average per day (note: not including sweetened tea/coffee)
* Known intolerance, sensitivity, or allergy to any ingredients in the study test products
* Self-reported pregnancy or breastfeeding or planning to become pregnant.
* Participation in any clinical trial within the past 30 days or any PepsiCo protocol within the past 6 months.
* Subjects who, in the opinion of the investigator, are unable or unlikely to comply with the dosing schedule and study evaluations.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in incremental area under the plasma glucose curve (ignoring area below the baseline, iAUC) over each 4-week intervention period | Before (-5 minutes and 0 minutes) and 15, 30, 45, 60, 90 and 120 minutes after overnight fasted subjects start to consume 50 grams of glucose on Day 1 and Day 29 of each of two 4-week intervention periods
  Finger stick blood samples obtained fasted prior to consuming 50 grams of glucose. Six additional finger stick blood samples obtained over the next 2 hours beginning 15 minutes after consumption.

SECONDARY OUTCOMES:
Fecal microbiota composition | Pre-dose baseline and Week 4 for each of two 4-week dosing periods
  Stool sample measured via 16S rRNA sequencing

OTHER OUTCOMES:
Fasting serum short-chain fatty acid (SCFA) | Pre-dose baseline Day 1 and Day 29 of each of two 4-week dosing periods
  Serum from venous blood sample
Fasting serum bile acids (BA) | Pre-dose baseline Day 1 and Day 29 of each of two 4-week dosing periods
  Serum from venous blood sample
Serum glucose total AUC 0-2 hours, peak concentrations and peak rises for glucose; glucose concentrations and increments at each time point over 2 hours | Fasted at -5 minutes Time 0 pre-dose, post-dose 15, 30, 45, 60, 90 and 120 minutes post-dose.
  Finger stick blood samples in unit mmol/L
Serum insulin iAUC 0-2 hours; total AUC 0-2 hours, peak concentrations and peak rises for insulin; insulin concentrations and increments at each time point over 2h | Fasted at -5 minutes, Time 0 pre-dose, post-dose 15, 30, 45, 60, 90 and 120 minutes post-dose.
  Finger stick blood samples in unit mU/L
Indices of insulin resistance | Pre-dose baseline Day 1 and Day 29 of each of two 4-week dosing periods
  Calculated from fasting plasma glucose (FPG) and fasting serum insulin (FSI) (HOMA-IR) (no units) = FPG(mmol/L) x FSI(mU/L)/22.5
Indices of insulin secretion | Pre-dose baseline Day 1 and Day 29 of each of two 4-week dosing periods
  Calculated from fasting plasma glucose and fasting serum insulin (HOMA-B ) (no units) = 20 x FSI(mU/L)/(FPG(mmol/L) - 3.5)
Matsuda's index of insulin sensitivity | Pre-dose baseline Day 1 and Day 29 of each of two 4-week dosing periods
  Derived from the plasma glucose and serum insulin concentrations measured during the oral glucose tolerance test (OGTT) (no units)
Abdul-Ghani et al. indices of liver insulin sensitivity | Pre-dose baseline Day 1 and Day 29 of each of two 4-week dosing periods, from 0-30 minutes after the oral glucose load for plasma glucose and serum insulin
  Total areas under the curve (no units), calculated as (gAUC0-30) x (iAUC0-30
Abdul-Ghani et al. indices of muscle insulin sensitivity | Pre-dose baseline Day 1 and Day 29 of each of two 4-week dosing periods, from 0-120 minutes
  Calculated as (dG/dt)/INS (no units)
Intake of dietary fiber and selected macro- and micro-nutrients | Recorded consumption for 2 weekdays and 1 weekend day during the week before the visit at the end of each 28 day dosing period
  Assessed using 3-day diet records
Optional Outcome: Glucagon-like peptide-1 (GLP-1) concentrations pending significant changes in butyrate concentrations | Pre-dose baseline Day 1 and Day 29 of each of two 4-week dosing periods
  Serum from venous blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — INQUIS Clinical Research
Locations (1):
- INQUIS Clinical Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No